CLINICAL TRIAL: NCT04102176
Title: HALT NUCs: Halting Nucleoside Analogue Therapy in Chronic Hepatitis B
Brief Title: Halting Nucleoside Analogues in Chronic Hepatitis B
Acronym: HALT-NUCS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seng Gee Lim (Other)
Collaborators: Tan Tock Seng Hospital (Other); Singapore General Hospital (Other); Changi General Hospital (Other)
Responsible Party: Sponsor-Investigator, Seng Gee Lim, Director of Hepatology, National University Health System, Singapore
Organization: National University Health System, Singapore (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIRG17may042
Record Dates: First submitted 2019-05-27; First posted 2019-09-25 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Chronic Hepatitis B
Keywords: chronic hepatitis B; nucleoside analogues; stopping; discontinuing
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Intervention Model Description: Parallel arm study randomised 1:2
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Continue nucleos(t)ide analogue (Active Comparator): patients will be given open label tenofovir alafenamide
  Interventions: Other: Continue nucleos(t)ide analogue
- Stopping nucleos(t)ide analogue (Experimental): patients will stop nucleos(t)ide therapy (such as entecavir, tenofovir, lamivudine or adefovir)
  Interventions: Other: stopping nucleos(t)ide therapy

INTERVENTIONS:
Other: stopping nucleos(t)ide therapy — patients taking nucleoside(t)ide therapy will stop treatment
  Arms: Stopping nucleos(t)ide analogue
Other: Continue nucleos(t)ide analogue — Continue nucleos(t)ide analogue
  Arms: Continue nucleos(t)ide analogue

SUMMARY:
Most patients with Chronic Hepatitis B are on nucleoside analogy (NA) long term, but this leads to HBsAg loss (defined as functional cure) of only 2% at 6 years. Recently a number of studies have shown significant HBsAg loss rates after stopping nucleoside analogues (NA). However, no criteria to select such patients have been evaluated. Consequently, the objective of the study is not only to determine the proportion of patients able to achieve HBsAg loss in those with qHBsAg≤100IU/ml. The study is designed as a randomised control trial with 1:2 parallel arm randomisation to continuing NA or stopping therapy. Patients will be monitored after stopping therapy for Hepatitis B flares and also to document HBsAg loss.

DETAILED DESCRIPTION:
Chronic Hepatitis B (CHB) affects over 250 million persons and is considered one of the major causes of mortality and morbidity globally. Standard treatment consists of nucleos(t)ide analogues (NA) or peginterferon (PEG). There has been increasing interested in HBsAg loss, defined as functional cure. However this has been difficult to achieve with NA, and although rates of HBsAg loss are higher with PEG, they are still <10%. However, a number of studies have shown that HBsAg loss rates were significantly higher in those who stopped NA. A study from Greece by Hadziyannis had a 39% HBsAg loss after patients stopped adefovir therapy. Further studies have shown similar results, and those not able to clear HBsAg have had quiescent disease, although some patients had to restart therapy usually due to hepatitis B flares. No deaths have been reported. Consequently, while stopping therapy has led to HBsAg loss in some patients, it is not clear which patients would benefit the most. The prior studies have indicated that patients most likely to lose HBsAg had low qHBsAg levels and a level ≤100 IU/ml had a high possibility of HBsAg loss. Consequently, we propose to test whether patients with CHB on NA >1year and without liver cirrhosis and with qHBsAg≤100 IU/ml are able to lose HBsAg compared to those who continue NA. The study is designed as a parallel arm RCT randomised 1:2 to continue NA versus stop NA. Patients will be monitored regularly for clinical status, virological markers, and liver markers. The primary endpoint is HBsAg loss at the end of the study in those who stop versus those who continue NA. Additional outcomes will be hepatitis B flares, inactive hepatitis B status, virological relapse, and restarting therapy.

ELIGIBILITY:
Inclusion Criteria:

* • Between 21 and 75 years old.

  * Documented to be HBsAg positive for ≥ 6 months.
  * On any NA (lamivudine, adefovir, entecavir, telbivudine tenofovir) for ≥ 1 year
  * HBV DNA <15 IU/ml at screening (undetectable)
  * Quantitative HBsAg <100 IU/ml
  * Patient has agreed not to take any other investigational drug or systemic anti-viral, cytotoxic, corticosteroid, immunomodulatory agents or Chinese traditional remedies unless clinically indicated.
  * Patient is able to give written consent prior to study start and to comply with the study requirements.
  * Women of childbearing age must have a negative serum (ß-HCG) pregnancy test taken with 14 days of starting therapy

Exclusion Criteria:

* • Evidence of liver cirrhosis based on liver biopsy, fibroscan score >10.5 kpa, or MRE score>5.5kpa, or clinical evidence of cirrhosis demonstrated by presence of esophageal varices, obvious features of cirrhosis on ultrasound within the last 12 months

  * Evidence of decompensated liver disease or hepatocellular carcinoma.
  * HIV antibody or HCV antibody or HDV antibody positivity
  * Creatinine > 1.5 times upper limit of normal
  * INR > 1.5, uncorrected by Vitamin K therapy.
  * Any interferon, Immunomodulators, systemic cytotoxic agents, or systemic corticosteroids within 6 months before trial entry.
  * Prolonged exposure to known hepatotoxins such as alcohol or drugs.
  * History of clinically relevant psychiatric disease, seizures, central nervous system dysfunction, severe pre-existing cardiac, renal, hematological disease or medical illness that in the investigator's opinion might interfere with therapy.
  * Malignant disease within 5 years of trial entry.
  * Women who are pregnant and who are not practicing adequate birth control measures, or who are lactating

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2019-01-29 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
HBsAg loss | Through year 3
  Absence of HBsAg by ELISA

SECONDARY OUTCOMES:
Hepatitis B flare | Through year 3
  increase in ALT associated with increase in HBV DNA
virological relapse | Through year 3
  increase in HBV DNA without increase in ALT
Restarting antiviral therapy | Through year 3
  Those who have to start therapy based on clinical indications after stopping therapy

CONTACTS AND LOCATIONS:
Overall Officials: Seng Gee Lim, MBBS MD, Principal Investigator — National University Health System
Locations (1):
- National University Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No